CLINICAL TRIAL: NCT05592925
Title: Association Between Multiple Coagulation-related Factors and Lymph Node Metastasis in Patients With Gastric Cancer: A Retrospective Cohort Study
Acronym: MA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Feng Tian, Director, Shandong Provincial Hospital
Other Study IDs: FTian
Record Dates: First submitted 2022-10-18; First posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Gastric Cancer Stage; Lymph Node Metastasis
Keywords: gastric cancer; lymph node metastasis; maximum amplitude; prognostic factor
MeSH Terms: conditions — Lymphatic Metastasis; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- N0: gastric cancer patients with no lymph node metastasis
  Interventions: Diagnostic Test: coagulation-related factors
- N+: gastric cancer patients with lymph node metastasis, including patients with N1, N2 and N3 stage cancer
  Interventions: Diagnostic Test: coagulation-related factors

INTERVENTIONS:
Diagnostic Test: coagulation-related factors — We retrospectively evaluated the relationship between lymph node metastasis and coagulation-related factors in 516 patients with T4a stage gastric cancer.

SUMMARY:
We initially selected a total of 1128 patients with primary gastric cancer who presented at Shandong Provincial Hospital between January 2018 and October 2022, and retrospectively collected their clinical and pathological data. And retrospectively analyzed preoperative baseline characteristics, preoperative laboratory tests, and postoperative pathological results for these patients

ELIGIBILITY:
Inclusion Criteria:

1. patients with primary gastric malignant tumors,
2. patients who underwent radical resection of gastric cancer,
3. patients with a postoperative pathology of adenocarcinoma or signet ring cell carcinoma according to the WTO pathological classification,

Exclusion Criteria:

1. patients who have distant metastases, such as liver or lung metastases, were found on preoperative ultrasound and computed tomography (CT) examinations,
2. patients who have received preoperative neoadjuvant chemotherapy,
3. patients who take anticoagulant drugs (such as aspirin) prior to surgery,
4. patients who had any previous coagulation disorder.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with primary gastric cancer
Sampling Method: Probability Sample
Enrollment: 516 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative coagulation-related factors (MA values) of patients | Three years
  MA values(mm). Measure the data of preoperative MA values in 516 gastric cancer patients to see wether this indicator correlated with tumor stage in patients with gastric cancer.
Preoperative coagulation-related factors (platelet counts) of patients | Three years
  Platelet counts（x10^9/L). Measure the data of preoperative platelet counts in 516 gastric cancer patients to see wether this indicator correlated with tumor stage in patients with gastric cancer.
Preoperative coagulation-related factors (fibrinogen levels) of patients | Three years
  Fibrinogen levels (g/L). Measure the data of preoperative fibrinogen levels in 516 gastric cancer patients to see wether this indicator correlated with tumor stage in patients with gastric cancer.
Preoperative coagulation-related factors (D-dimer) of patients | Three years
  D-dimer (mg/L). Measure the data of preoperative D-dimer in 516 gastric cancer patients to see wether this indicator correlated with tumor stage in patients with gastric cancer.
Postoperative pathological results of tumor T stage. | Three years
  Recording the postoperative pathological tumor T stage in 516 patients with gastric cancer.
Postoperative pathological results of tumor N stage. | Three years.
  Recording the postoperative pathological tumor N stage in 516 patients with gastric cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Tian, Doctor, Principal Investigator — Shandong Provincial Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
After the article is published, the original data can be obtained by contacting the project leader.